CLINICAL TRIAL: NCT01938612
Title: A Phase I, Open-Label, Multicentre Study to Evaluate the Safety, Tolerability and Pharmacokinetics of MEDI4736 in Patients With Advanced Solid Tumours
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D4190C00002
Record Dates: First submitted 2013-09-05; First posted 2013-09-10 (Estimated); Last update posted 2021-03-12 (Actual); Status verified 2021-03

CONDITIONS: Advanced Solid Tumors
Keywords: MEDI4736; Advanced solid tumors; squamous cell carcinoma of the head and Neck; biliary tract cancer; squamous cell carcinoma of esophagus cancer; B7-H1; PD-L1
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Biliary Tract Neoplasms | interventions — durvalumab; tremelimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- MEDI4736 Q2W (Experimental): Evaluate MEDI4736 given every 2 weeks
  Interventions: Drug: MEDI4736
- MEDI4736 Q3W (Experimental): Evaluate MEDI4736 given every 3 weeks
  Interventions: Drug: MEDI4736
- MEDI4736 Dose Expansion (Experimental): evaluate MEDI4736 given every 2 weeks
  Interventions: Drug: MEDI4736
- MEDI4736 Q4W (Experimental): Evaluate MEDI4736 given every 4 weeks
  Interventions: Drug: MEDI4736
- MEDI4736 combined with another drug (Experimental): evaluate MEDI4736 in combination with another drug given every 4 weeks
  Interventions: Drug: tremelimumab

INTERVENTIONS:
Drug: MEDI4736 — MEDI4736 will be administered by IV infusion every 14, 21 or 28 days.
  Arms: MEDI4736 Dose Expansion; MEDI4736 Q2W; MEDI4736 Q3W; MEDI4736 Q4W
Drug: tremelimumab — tremelimumab is administered by IV infusion every 4 weeks
  Arms: MEDI4736 combined with another drug

SUMMARY:
This is a phase I, open-label, multicentre study of MEDI4736 administered intravenously with a standard 3+3 dose-escalation phase to evaluate safety, tolerability, and pharmacokinetics in patients with advanced solid tumor followed by an expansion phase in patients with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* In the dose-escalation phase: patients with advanced solid tumors refractory to standard treatment, intolerant of standard treatment, or for which no standard therapy exists.

In the dose-expansion phase: histologically- or cytologically-confirmed advanced or metastatic biliary tract cancer (BTC), esophagus cancer(EC) (squamous cell carcinoma) or squamous cell carcinoma of the head and neck (SCCHN). - men or women. - Eastern Cooperative Oncology Group (ECOG) status of 0 or 1. - Adequate organ and marrow function. - Subjects must have at least 1 measurable lesion. - Available archived tumor tissue sample. - Willingness to provide consent for biopsy samples.

Exclusion Criteria:

* Any prior Grade ≥ 3 irAE while receiving immunotherapy - Prior exposure to any anti-PD-1 or anti-PD-L1 antibody - Active or prior documented autoimmune disease within the past 2 years - History of primary immunodeficiency - Symptomatic or untreated central nervous system (CNS) metastases requiring concurrent treatment - Women who are pregnant or lactating - Uncontrolled intercurrent illness - Known history of tuberculosis - Known to be human immunodeficiency virus (HIV) positive - Hepatitis B or C infection - Other invasive malignancy within 5 years

Ages: 20 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 269 (Actual)
Dates: Start 2013-09-12 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2020-11-25 (Actual)

PRIMARY OUTCOMES:
Number of participants experiencing dose-limiting toxicities, adverse events (AEs), serious adverse events (SAEs) | 90 days after the last dose of MEDI4736
  Safety profile will be assessed through number of participants experiencing adverse events (AEs), serious adverse events (SAEs), laboratory evaluations, vital signs, and physical examinations.

SECONDARY OUTCOMES:
Area under the concentration of MEDI4736 time curve | Up to 90 days after the last dose of MEDI4736
  If data allow, noncompartmental PK parameter (AUC) will be estimated.
Percentage of participants who developed detectable anti-drug antibodies (ADAs). | Up to 6 months after the last dose of MEDI4736 or up to 1 month after the last dose of tremelimumab where applicable.
  The immunogenic potential of MEDI4736 or tremelimumab will be assessed by summarizing the number percentage of subjects who develop detectable anti-drug antibodies (ADAs).
Objective response rate (ORR) | From first dose of study drug until death or up to 2 years
Maximum tolerated dose (MTD) or optimal biological dose (OBD) | 90 days after the last dose of MEDI4736
  maximum tolerated dose (MTD) or optimal biological dose (OBD) of MEDI4736, if possible
Maximum concentration of MEDI4736 | Up to 90 days after the last dose of MEDI4736
  If data allow, noncompartmental PK parameter (Cmax) will be estimated.
Clearance | Up to 90 days after the last dose of MEDI4736
  If data allow, noncompartmental PK parameter (CL) will be estimated.
half-life after administration of MEDI4736 | Up to 90 days after the last dose of MEDI4736
  If data allow, noncompartmental PK parameter (t½) will be estimated.
Disease control rate (DCR) | From first dose of study drug until death or up to 2 years
Duration of response (DoR) | From first dose of study drug until death or up to 2 years
Progression-free survival (PFS) | From first dose of study drug until death or up to 2 years
  Alive and progression free at 6 months (APF6) and 12 months (APF12) will be obtained using the Kaplan-Meier plot of PFS.
Overall survival (OS) | From first dose of study drug until death or up to 2 years
  The proportion of patients alive at 12 months will be obtained from the Kaplan-Meier plot of OS.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Iannone, MD, Study Director — AstraZeneca
Locations (19):
- Japan (15):
  - Research Site, Beppu-shi
  - Research Site, Chūōku
  - Research Site, Kashiwa
  - Research Site, Kitaadachi-gun
  - Research Site, Kōtoku
  - Research Site, Kure-shi
  - Research Site, Matsuyama
  - Research Site, Nagoya
  - Research Site, Osaka
  - Research Site, Sapporo
  - Research Site, Sayama
  - Research Site, Suita-shi
  - Research Site, Sunto-gun
  - Research Site, Takatsuki-shi
  - Research Site, Yokohama
- Research Site, Seoul, South Korea
- Taiwan (3):
  - Research Site, Tainan
  - Research Site, Taipei
  - Research Site, Taoyuan District

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Doki Y, Ueno M, Hsu CH, Oh DY, Park K, Yamamoto N, Ioka T, Hara H, Hayama M, Nii M, Komuro K, Sugimoto M, Tahara M. Tolerability and efficacy of durvalumab, either as monotherapy or in combination with tremelimumab, in patients from Asia with advanced biliary tract, esophageal, or head-and-neck cancer. Cancer Med. 2022 Jul;11(13):2550-2560. doi: 10.1002/cam4.4593. Epub 2022 May 24. PMID 35611499